CLINICAL TRIAL: NCT02604264
Title: Product Evaluation for the Effectiveness of the ClearGuard™ HD End Cap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pursuit Vascular, Inc. (Industry)
Collaborators: Fresenius Medical Care North America (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLP-0001
Record Dates: First submitted 2015-11-11; First posted 2015-11-13 (Estimated); Results first posted 2017-05-01 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-06

CONDITIONS: End Stage Renal Disease (ESRD)
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ClearGuard HD end cap (Active Comparator): Treatment
  Interventions: Device: ClearGuard HD end cap
- Standard hemodialysis end cap (No Intervention): Control

INTERVENTIONS:
Device: ClearGuard HD end cap — The ClearGuard HD End Cap elutes chlorhexidine acetate into the hemodialysis catheter hub
  Arms: ClearGuard HD end cap

SUMMARY:
To assess positive blood cultures (PBCs) in hemodialysis central venous catheter (CVC) patients using two FDA cleared devices: ClearGuard HD end caps compared to conventional end caps.

ELIGIBILITY:
Inclusion Criteria:

* All patients dialyzing with a central venous catheter

Exclusion Criteria:

* Known allergy to chlorhexidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2912 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Hymes, MD, Principal Investigator — Fresenius Medical Care North America
Locations (1):
- Frenova Renal Research, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hymes JL, Mooney A, Van Zandt C, Lynch L, Ziebol R, Killion D. Dialysis Catheter-Related Bloodstream Infections: A Cluster-Randomized Trial of the ClearGuard HD Antimicrobial Barrier Cap. Am J Kidney Dis. 2017 Feb;69(2):220-227. doi: 10.1053/j.ajkd.2016.09.014. Epub 2016 Nov 10. PMID 27839894
- [Derived] Almeida BM, Moreno DH, Vasconcelos V, Cacione DG. Interventions for treating catheter-related bloodstream infections in people receiving maintenance haemodialysis. Cochrane Database Syst Rev. 2022 Apr 1;4(4):CD013554. doi: 10.1002/14651858.CD013554.pub2. PMID 35363884
- See also: Pursuit Vascular website — http://www.pursuitvascular.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: ClearGuard HD end cap: The ClearGuard HD End Cap elutes chlorhexidine acetate into the hemodialysis catheter hub
- Control: Standard hemodialysis end cap
Period: Run-In
Arm/Group | Treatment | Control
Started (The 1-mo run-in period data was used to determine pre-study demographics and PBC rate.) | 618 | 611 (The 1-mo run-in period data was used to determine pre-study demographics and PBC rate.)
Completed | 618 | 611
Not Completed | 0 | 0
Period: Intervention
Arm/Group | Treatment | Control
Started | 1445 | 1467
Completed | 1245 | 1225
Not Completed | 200 | 242
Not completed — Didn't use CVC for at least 21 days | 200 | 242

BASELINE CHARACTERISTICS:
Population: This is the intervention population data. The baseline data came from the 1 month run-in period prior to the start of the intervention period and is referred to as the run-in rather than baseline period. The run-in data was used to determine pre-study demographics and PBC rate.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 1245 | 1225 | 2470
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (15.1) | 60.6 (15.1) | 61.1 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 591 | 559 | 1150
  Male | 654 | 666 | 1320
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 24 | 25
  Asian | 13 | 12 | 25
  Native Hawaiian or Other Pacific Islander | 3 | 4 | 7
  Black or African American | 566 | 495 | 1061
  White | 609 | 631 | 1240
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 53 | 59 | 112
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1245 | 1225 | 2470

OUTCOME MEASURES:

1. Primary Outcome: Positive Blood Cultures (PBCs) Per 1,000 Central Venous Catheter (CVC)-Days
Description: This was calculated by dividing the cumulative number of PBCs by cumulative time at-risk as follows.
  The National Healthcare Safety Network (NHSN) Center for Disease Control (CDC) 21-day outpatient hemodialysis patient rule is as follows: A PBC is considered a new event and counted only if it occurred 21 days or more after a previously reported PBC in the same patient; new PBC events are based on blood cultures drawn as an outpatient or within one calendar day after a hospital admission. Following a PBC additional same-type events were counted beginning 21 days following the initial event; the CVC-days were counted during this period. The CVC-days were calculated by summing the number of days each patient was at-risk of accruing a PBC. This analysis included all subjects that participated in the study that were not otherwise censored to more accurately count CVC-days.
Time Frame: Up to 12 months
Measure: Number; unit: PBCs per 1,000 CVC-days
Arm/Group | Treatment | Control
Number analyzed (Participants) | 1245 | 1225
PBCs per 1,000 CVC-days | 0.26 | 0.59

ADVERSE EVENTS:
Time Frame: 1 year
Description: The run-in data was used to determine pre-study demographics and PBC rate so no adverse event analysis was performed for the this period. This was a pragmatic post market study. There was an informed consent waiver and there were no study case report forms (CRF's). Treatment arm adverse events were monitored during the 12-month intervention period using the FDA Manufacturer and User Facility Device Experience (MAUDE) database and none were reported.
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 134/1245 | 127/1225
Serious Adverse Events (participants affected / at risk) | 0/1245 | 0/1225
Other Adverse Events (participants affected / at risk) | 0/1245 | 0/1225

LIMITATIONS AND CAVEATS:
This was a pragmatic post market study. There was an informed consent waiver and no CRF's. Treatment arm adverse events during the 12-month intervention period were monitored using the FDA MAUDE database and none were reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No